CLINICAL TRIAL: NCT00130117
Title: Randomized, Double-blind, Placebo-controlled Trial of Human Recombinant Leptin (r-metHuLeptin) for the Treatment of Hypothalamic (Exercise-Induced) Amenorrhea
Brief Title: Study of Leptin for the Treatment of Hypothalamic Amenorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Research Resources (NCRR) (NIH); Amgen (Industry)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004P000123; 1R34HD048526-01 (NIH); 5M01RR001032-32 (NIH)
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Amenorrhea
Keywords: leptin; hypothalamic amenorrhea; exercise-induced amenorrhea; neuroendocrine function; bone metabolism
MeSH Terms: conditions — Amenorrhea | interventions — recombinant methionyl human leptin; metreleptin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- r-metHuLeptin (Experimental): r-metHuLeptin administered subcutaneously.
  Interventions: Drug: r-metHuLeptin; Drug: Oral Contraceptive Pills (OCPs)
- Oral Contraceptive Pills (OCPs) (Placebo Comparator): PLACEBO
  Interventions: Drug: Oral Contraceptive Pills (OCPs); Other: Placebo

INTERVENTIONS:
Drug: r-metHuLeptin — Starting dose: 0.08mg/kg once daily Subcutaneous injection.
  Other Names: metreleptin
  Arms: r-metHuLeptin
Drug: Oral Contraceptive Pills (OCPs) — Sprintec taken orally once daily.
  Other Names: OCPs
Other: Placebo — placebo (no active medication)
  Arms: Oral Contraceptive Pills (OCPs)

SUMMARY:
The purpose of this study is to determine whether administration of an investigational medication called leptin (r-metHuLeptin) in replacement doses can improve bone health, reproductive function, hormone levels, immune function, and overall sense of well-being in women with hypothalamic (exercise-induced) amenorrhea (HA) who are being treated with oral contraceptive pills (OCPs), compared to placebo. Women with hypothalamic amenorrhea have low leptin levels. This study is based on the hypothesis that the relative leptin deficiency in women with hypothalamic (exercise-induced) amenorrhea may be the reason for the lack of menstrual cycles, hormone abnormalities, and bone loss associated with this condition.

DETAILED DESCRIPTION:
Leptin is a hormone secreted by fat cells under normal conditions and acts in the brain to regulate energy usage and hormone levels. Women with HA who do not have regular periods have low leptin levels and may also have other hormone abnormalities as well as loss of bone density (osteopenia or osteoporosis). This study will evaluate how leptin (a fat cell hormone that normally circulates in the blood) affects bone density, menstrual periods, hormone levels, bone metabolism (how bone forms and turns over), immune function (how well the body can fight infection), metabolic rate (how many calories are used at rest), and overall sense of well-being and appetite in women with HA (i.e. no regular menstrual periods due to low levels of pituitary hormones that regulate estrogen production from the ovary). It will also investigate whether leptin replacement can be used as an adjunct to the current standard of care for HA patients, i.e. OCPs.

Part A is a Randomized, placebo-controlled 36-week study. Part B is an Optional open-label 52-week study. There will also be an optional Reward Sub-study, including healthy controls, designed to investigate leptin's relation to reward processing by collecting participants' brain and behavioral responses to images (e.g., pictures of food vs. non-food). Brain responses will be collected and will also be assessed via functional Magnetic Resonance Imaging (fMRI).

Comparison: Part A = leptin-treated group to placebo-treated group and Part B optional sub study = leptin-treated group to health controls

ELIGIBILITY:
Inclusion criteria for HA subjects

* Hypothalamic amenorrhea of at least 6 months duration with low or normal LH and FSH, e.g. due to strenuous exercise (running >20 miles per week or equivalent) or low weight
* Can be secondary HA OR primary HA with some pubertal development and normal screening labs
* Age 18-35 years old
* Body weight within +/- 15% of ideal body weight and stable for 6 months (no change > 5 lbs)
* Baseline leptin <5 ng/mL (except for the Cognitive Sub-Study Baseline visit where baseline leptin will be greater than 5ng/mL)

Inclusion criteria for eumenorrheic controls for Reward Sub-study

* Normal menstrual cycles (between 25 and 35 days)
* Age 18-35
* Body weight within +/- 15% of ideal body weight and stable 6 months (no change > 5 lbs)
* Baseline leptin >5 ng/mL

Exclusion criteria:

* We will exclude subjects with:
* Significant medical history that may affect the concentrations of the hormones to studied or ability to participate in the study
* renal or hepatic disease (creatinine > 1.4, AST/ALT > 2x upper limit of normal)
* diagnosed diabetes mellitus
* myocardial ischemia
* malignancy (other than basal cell carcinoma of the skin or in situ carcinoma of the cervix)
* malabsorption
* alcoholism, drug abuse, or smoking
* active eating disorder
* depression or other psychiatric disease
* anemia (Hb10 gm/dL on 2 occasions)
* Conditions that are contraindicated for oral contraceptive use:
* Thrombophlebitis or thromboembolic disorders
* A past history of deep vein thrombophlebitis or thromboembolic disorders
* Cerebral vascular or coronary artery disease
* Known or suspected carcinoma of the breast
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Hepatic adenomas or carcinomas
* Cholestatic jaundice of pregnancy or jaundice with prior OCP use
* Other endocrine causes of amenorrhea, e.g.
* hyperprolactinemia
* hypothyroidism or hyperthyroidism
* Cushing's syndrome
* congenital adrenal hyperplasia (elevated 17 OH progesterone)
* polycystic ovarian syndrome (elevated androgens or LH/FSH ratio >1.5)
* primary ovarian failure (elevated FSH)
* On medications known to affect the hormones to be measured such as
* glucocorticoids
* anti seizure medications
* thyroid hormones
* estrogen (must be off at least 3 months prior to participating in the study)
* A known history of anaphylaxis or anaphylactoid-like reactions, or a known hypersensitivity to E. Coli derived proteins
* Breast feeding, pregnant, or wanting to become pregnant during the next 6 months.
* We will screen for these conditions through a detailed history and systems review, physical examination, laboratory evaluation (as described above in Screening Methods), and EKG.
* In the Reward Sub-study subjects will be asked to fill out a standard BIDMC MRI safety screening form prior to entering the magnet.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD, ScD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center General Clinical Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Welt CK, Chan JL, Bullen J, Murphy R, Smith P, DePaoli AM, Karalis A, Mantzoros CS. Recombinant human leptin in women with hypothalamic amenorrhea. N Engl J Med. 2004 Sep 2;351(10):987-97. doi: 10.1056/NEJMoa040388. PMID 15342807
- [Background] Mantzoros CS, Magkos F, Brinkoetter M, Sienkiewicz E, Dardeno TA, Kim SY, Hamnvik OP, Koniaris A. Leptin in human physiology and pathophysiology. Am J Physiol Endocrinol Metab. 2011 Oct;301(4):E567-84. doi: 10.1152/ajpendo.00315.2011. Epub 2011 Jul 26. PMID 21791620
- [Result] Sienkiewicz E, Magkos F, Aronis KN, Brinkoetter M, Chamberland JP, Chou S, Arampatzi KM, Gao C, Koniaris A, Mantzoros CS. Long-term metreleptin treatment increases bone mineral density and content at the lumbar spine of lean hypoleptinemic women. Metabolism. 2011 Sep;60(9):1211-21. doi: 10.1016/j.metabol.2011.05.016. Epub 2011 Jul 7. PMID 21741057
- [Result] Chou SH, Chamberland JP, Liu X, Matarese G, Gao C, Stefanakis R, Brinkoetter MT, Gong H, Arampatzi K, Mantzoros CS. Leptin is an effective treatment for hypothalamic amenorrhea. Proc Natl Acad Sci U S A. 2011 Apr 19;108(16):6585-90. doi: 10.1073/pnas.1015674108. Epub 2011 Apr 4. PMID 21464293
- [Derived] Chrysafi P, Perakakis N, Farr OM, Stefanakis K, Peradze N, Sala-Vila A, Mantzoros CS. Leptin alters energy intake and fat mass but not energy expenditure in lean subjects. Nat Commun. 2020 Oct 13;11(1):5145. doi: 10.1038/s41467-020-18885-9. PMID 33051459
- [Derived] Bouzoni E, Perakakis N, Mantzoros CS. Circulating profile of Activin-Follistatin-Inhibin Axis in women with hypothalamic amenorrhea in response to leptin treatment. Metabolism. 2020 Dec;113:154392. doi: 10.1016/j.metabol.2020.154392. Epub 2020 Oct 10. PMID 33045195
- [Derived] Foo JP, Polyzos SA, Anastasilakis AD, Chou S, Mantzoros CS. The effect of leptin replacement on parathyroid hormone, RANKL-osteoprotegerin axis, and Wnt inhibitors in young women with hypothalamic amenorrhea. J Clin Endocrinol Metab. 2014 Nov;99(11):E2252-8. doi: 10.1210/jc.2014-2491. Epub 2014 Aug 22. PMID 25148234
- [Derived] Hwang JJ, Thakkar B, Chamberland JP, Mantzoros CS. Circulating fetuin-A levels are not affected by short and long-term energy deprivation and/or by leptin administration. Metabolism. 2014 Jun;63(6):754-9. doi: 10.1016/j.metabol.2014.02.006. Epub 2014 Feb 17. PMID 24703486
- [Derived] Matarese G, La Rocca C, Moon HS, Huh JY, Brinkoetter MT, Chou S, Perna F, Greco D, Kilim HP, Gao C, Arampatzi K, Wang Z, Mantzoros CS. Selective capacity of metreleptin administration to reconstitute CD4+ T-cell number in females with acquired hypoleptinemia. Proc Natl Acad Sci U S A. 2013 Feb 26;110(9):E818-27. doi: 10.1073/pnas.1214554110. Epub 2013 Feb 4. PMID 23382191
- [Derived] Aronis KN, Diakopoulos KN, Fiorenza CG, Chamberland JP, Mantzoros CS. Leptin administered in physiological or pharmacological doses does not regulate circulating angiogenesis factors in humans. Diabetologia. 2011 Sep;54(9):2358-67. doi: 10.1007/s00125-011-2201-x. Epub 2011 Jun 10. PMID 21660636
- [Derived] Alonso-Alonso M, Ziemke F, Magkos F, Barrios FA, Brinkoetter M, Boyd I, Rifkin-Graboi A, Yannakoulia M, Rojas R, Pascual-Leone A, Mantzoros CS. Brain responses to food images during the early and late follicular phase of the menstrual cycle in healthy young women: relation to fasting and feeding. Am J Clin Nutr. 2011 Aug;94(2):377-84. doi: 10.3945/ajcn.110.010736. Epub 2011 May 18. PMID 21593494
- See also: Click here for more information about the Mantzoros Research Group. — http://www.bidmc.org/Research/Departments/Medicine/Divisions/Endocrinology/Laboratories/MantzorosLab.aspx
- See also: Click here for more information about Beth Israel Deaconess Medical Center. — http://www.bidmc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo
  Oral Contraceptive Pills (OCPs): Sprintec taken orally once daily.
  Placebo: placebo (no active medication)
Period: Overall Study
Arm/Group | r-metHuLeptin | Placebo
Started | 11 | 9
Completed | 7 | 6
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | r-metHuLeptin | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (1.4) | 25.4 (1.2) | 26 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: the Difference Between the Placebo and Leptin Treated Groups in the Change in Bone Mineral Content(BMC) at the Anteroposterior (AP) Spine From Baseline to 36 Weeks
Time Frame: 36 weeks
Measure: Mean (Full Range); unit: g
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 7 | 6
g | 51.0 [43.4 to 58.2] | 58.2 [55.2 to 61.4]
Statistical Analysis 1: Comparison: r-metHuLeptin vs Placebo; Test type: Superiority or Other; p = 0.024, ANOVA
Statistical Analysis 2: Comparison: r-metHuLeptin vs Placebo; Test type: Superiority; p = 0.049, ANOVA

2. Secondary Outcome: Bone Markers - Ctx and Sclerostin
Time Frame: 36 weeks
Population: Only for subjects participating in both phase A and phase B (n=4), bone markers were assessed to see the change over 24 month period. All these patient got metreleptin treatment
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | r-metHuLeptin
Number analyzed (Participants) | 4
ng/mL
  CTX | 0.60 [0.39 to 0.83]
  Sclerostin | 0.08 [0.07 to 0.09]
Statistical Analysis 1: Comparison: r-metHuLeptin; Test type: Superiority or Other; p = 0.02, ANOVA — p value reflects treatment of leptin for "on-treatment", n=4; Median Difference (Final Values) = 0.60

3. Secondary Outcome: Body Composition BMI
Time Frame: 36 weeks
Measure: Mean (Standard Error); unit: BMI-kg/m^2
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 7 | 6
BMI-kg/m^2 | 20.8 (0.6) | 21.1 (0.6)

4. Secondary Outcome: Total Body BMD
Time Frame: 36 weeks
Measure: Median (Inter-Quartile Range); unit: g/cm^2
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 7 | 6
g/cm^2 | 1.07 [1.05 to 1.16] | 1.13 [1.09 to 1.23]

5. Secondary Outcome: Body Fat
Time Frame: 36 weeks
Measure: Mean (Standard Error); unit: fat %
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 7 | 6
fat % | 23.9 (1.4) | 20.8 (1.3)

6. Secondary Outcome: Total Body BMD
Time Frame: 9 months
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | r-metHuLeptin | Oral Contraceptive Pills (OCPs)
Number analyzed (Participants) | 10 | 9
g/cm2 | 1.09 [1.06 to 1.15] | 1.13 [1.10 to 1.23]

7. Secondary Outcome: Lumbar BMD
Time Frame: 9 months
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 10 | 9
g/cm2 | 0.92 [0.80 to 1.03] | 0.97 [0.90 to 1.01]

8. Secondary Outcome: Radial BMD
Time Frame: 9 months
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 10 | 9
g/cm2 | 0.54 [0.52 to 0.60] | 0.54 [0.53 to 0.56]

9. Secondary Outcome: Hip BMD
Time Frame: 9months
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | r-metHuLeptin | Placebo
Number analyzed (Participants) | 10 | 9
g/cm2 | 0.89 [0.80 to 1.03] | 0.88 [0.80 to 1.02]

ADVERSE EVENTS:
Description: 11 participants started on the metreleptin arm , although only 7 finished the study. hence participants at risk are 11
Arm/Group | r-metHuLeptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 2/11 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | r-metHuLeptin (N=11) | Placebo (N=6)
local injection site reactions with erythematous rashes (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Number of participants was small and, therefore, our observations need to be validated in studies with larger sample sizes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No